CLINICAL TRIAL: NCT06714825
Title: Phase 1 Single and Multiple Ascending Dose Study in Males and Females Assessing the Pharmacokinetics, Safety, and Pharmacodynamics of HS235 in Overweight and Obese Otherwise Healthy Subjects
Brief Title: Study of HS235 for Assessing the Pharmacokinetics, Safety, and Pharmacodynamics in Overweight/Obese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 35Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HS235-001
Record Dates: First submitted 2024-11-27; First posted 2024-12-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2024-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Product (Experimental): HS235 Subcutaneous Injection
  Interventions: Biological: HS235
- Placebo (Placebo Comparator): Subcutaneous Injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: HS235 — Up to 4 Single and 3 Multiple Ascending Doses
  Arms: Investigational Product
Drug: Placebo — Subcutaneous Injection
  Arms: Placebo

SUMMARY:
Study of HS235 for Assessing the Pharmacokinetics, Safety, and Pharmacodynamics of HS235 in Overweight and Obese Otherwise Healthy Subjects

DETAILED DESCRIPTION:
A Phase 1 Study Assessing the Pharmacokinetics, Safety, and Pharmacodynamics of HS235 in Overweight and Obese Otherwise Healthy Subjects: Single Ascending Dose (SAD) in Males and Postmenopausal Females and Multiple Ascending Dose (MAD) in Males and Females of Non-childbearing Potential

ELIGIBILITY:
Inclusion Criteria:

1. Male or female above 40 years of age, inclusive.
2. Body Mass Index (BMI) between 28 and 40 kg/m2, inclusive.
3. Body weight at or below 140 kg with a stable body weight.
4. In good health or with no clinically significant medical conditions
5. Females who are post-menopausal or are of Non-child bearing Potential.
6. Male subjects must be willing not to donate sperm for 90 days after the last dose.
7. Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria:

1. Females with a positive pregnancy test or who are lactating.
2. Subjects with diabetes or have previous history of diabetes.
3. Subjects who have recently donated blood, plasma and platelets.
4. Subjects with history of alcoholism or drug abuse.
5. Subjects who received systemic or topical medications, depot injections or implants, hormone replacement, non-prescribed medication or herbal remedies, or daily glucocorticoids for > 1 month in previous year.
6. Subjects with clinically significant abnormal pulse or blood pressure or temperature.
7. Subjects with a history of a clinically significant medical disorder or lab abnormality.
8. Subjects with a significant history of multiple drug allergies, including infusion reactions and hypersensitivity to any of the excipients of HS235.
9. Subjects who are carriers of the hepatitis B surface antigen (HBsAg) and are carriers of the hepatitis C antibody (except if Polymerase Chain Reaction Ribonucleic acid (PCR RNA) is negative); or have a positive result to the test for human immunodeficiency virus (HIV) antigen or antibody.
10. Subjects who have, in the opinion of the Investigator, an abnormality in the echocardiogram or 12-lead ECG that put them at increased risk during the study.
11. Current or history of treatment with medications that may cause significant weight gain or loss, within 3 months or 5 half-lives of screening.
12. Obesity induced by other endocrine disorders.
13. Previous surgical treatment for obesity.
14. Current or history of treatment with medications that may cause significant weight gain or loss.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence and Number of Adverse Events (AEs) | up to 106 days for Single dose and 147 days for multiple doses
  An AE is any untoward medical occurrence in a patient or clinical trial patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.The incidence and number of patients who experience an AE will be reported.

SECONDARY OUTCOMES:
Area under concentration time curve (AUC) zero to t | up to 106 days for Single dose and 147 days for multiple doses
  Blood samples will be collected to determine the Area under the concentration-time curve from time zero until the last observed concentration
Area under concentration time curve (AUC) zero-infinity | up to 106 days for Single dose and 147 days for multiple doses
  Blood samples will be collected to determine the Area under the concentration-time curve from time zero to infinity (extrapolated)
Maximum observed Plasma Concentration (Cmax) | up to 106 days for Single dose and 147 days for multiple doses
  Blood samples will be collected to determine Cmax
Time to maximum concentration (Tmax) | up to 106 days for Single dose and 147 days for multiple doses
  Blood samples will be collected to determine Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Monique Champagne, M.Sc., Study Director — VP, Clinical Operations
Locations (1):
- Syneos Clinical Research Unit, Québec, Quebec, Canada